CLINICAL TRIAL: NCT01531062
Title: Effect of Nigella Sativa on Lipid Profiles in Elderly: a Randomized Double-blinded Clinical Trial
Brief Title: Effect of Nigella Sativa on Lipid Profiles in Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Jimmy Tandradynata, Dr., Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nigella sativa
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Dyslipidemia
Keywords: nigella sativa; dyslipidemia; elderly
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nigella sativa (Experimental): Nigella sativa extracts, 300 mg twice daily
  Interventions: Drug: Nigella sative
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: black sticky rice

INTERVENTIONS:
Drug: Nigella sative — Nigella sativa seed extracts, 300 mg capsule bid, for 56 days
  Arms: Nigella sativa
Dietary Supplement: black sticky rice — 300 mg capsule bid, 56 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Nigella sativa seed extracts are effective in the treatment of dyslipidemia in elderly.

DETAILED DESCRIPTION:
Cardiovascular diseases are still common health problems worldwide. They are major causes of morbidity and mortality in many countries. Dyslipidemia is the main risk factor of cardiovascular events. Despite the invention of many conventional hypolipidemic drugs, the use of traditional medicine remains high, especially in elderly patients. However, evidence of the effectiveness of many herbs or other traditional drugs is lacking. Nigella sativa or black seeds are traditional herbs used for years in Middle East and India. They are believed to cure many diseases, including dyslipidemia. Therefore, a study is needed to prove their effectiveness as their use might improve our strategy to improve patients' compliance.

ELIGIBILITY:
Inclusion Criteria:

* age of 60 years or more
* having dyslipidemia (total cholesterol >200 mg/dL or LDL >100 mg/dL or triglyceride > 150 mg/dL or HDL < 40 mg/dL (male) or HDL < 50 mg/dL (female)

Exclusion Criteria:

* ALT or AST are two times of upper normal limit
* creatinine clearance test is below 30

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Decreased level of total cholesterol, LDL, dan triglyceride, and increased level of HDL | 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine Department, Faculty of Medicine, University Indonesia, Jakarta, Jakarta Special Capital Region, Indonesia